CLINICAL TRIAL: NCT07071831
Title: RetroPerc®-A Prospective, Multi-institutional Trial of Efficacy of the RetroPerc Device
Brief Title: RETRO Study (RETrograde Renal Access Outcomes)
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: RetroPerc Inc (Unknown)
Responsible Party: Principal Investigator, Bristol Whiles, MD, Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY00160854
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Renal Stones
Keywords: kidney stones
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous Nephrolithotomy: Participants with a single renal stone or total sum of 1.5 to 3 cm in maximum dimension of multiple stones undergoing percutaneous nephrolithotomy as part of their routine medical care using the RetroPerc® system to obtain renal access.
  Interventions: Device: RetroPerc®

INTERVENTIONS:
Device: RetroPerc® — The RetroPerc® will be used to obtain renal access.

SUMMARY:
The goal of this observational study is to learn about the benefit of using RetroPerc® in obtaining renal access for percutaneous nephrolithotomy. The device is already used in routine clinical practice by urologists around the country.

Participants who are already scheduled to undergo percutaneous nephrolithotomy as part of their regular care will be asked to participate.

DETAILED DESCRIPTION:
Retrograde nephrostomy access is well established as a safe method for nephrostomy creation and thus this study aims to perform a standard of care study. The device is already available, on the shelf, and used in routine clinical care. However, the study aims to take a closer look in a prospective fashion at this access technique to better understand specific variables that are not available on retrospective review of cases that have already undergone PCNL with this technique.

ELIGIBILITY:
Inclusion Criteria:

* Renal stone or total linear sum of 1.5-3cm cm in maximum dimension (largest diameter in axial or coronal)--- multiple stones should be summed to determine stone size.
* Age >=18 years of age
* Gender: both men and women included.
* Ethnic background: all ethnicities will be included in the study population and the specific ethnic diversity present in the study population will reflect the geographic distributions of the participating institutions.
* Plan for PCNL in the supine position

Exclusion Criteria:

* Active pregnancy
* BMI >45
* Severe Hydronephrosis - renal pelvis diameter > 20mm
* Flank window < 4 cm are ineligible for puncture
* Previous ipsilateral PCNL
* Currently with "useful" nephrostomy tube on ipsilateral side
* Uncorrectable coagulopathies
* Untreated urinary tract infection
* Subjects with significant morbidities such as American Society of Anesthesiologists (ASA) score ≥ 4, severe spinal cord injuries, severe cardiopulmonary insufficiency, uncontrolled diabetes, neurological disorders, bedbound, anticipated life expectancy less than 5 years, or any other comorbidity, that in the opinion of the principal investigator could represent an increased peri-operative risk for the subject;
* Ipsilateral partial nephrectomy
* History of ipsilateral ureteral reimplantation or ureteral reconstruction;
* History of Simple or radical prostatectomy
* History of cystectomy
* History of calyceal diverticula stone;
* History of renal donation or transplant;
* Any other previous pelvic surgical treatment that could put the subject at greater procedural complication risk or technical difficulty;
* Ureteral ipsilateral stricture, untreated;
* Ureteral stricture, untreated (not to include "tight" ureter);
* Any other bladder, ureteral or kidney congenital genitourinary abnormalities (e.g. Horseshoe kidney, ipsilateral duplicated or partially duplicated collecting system, ipsilateral ectopic kidney, cross-fused ectopia, bifid renal pelvis with no horizontally directed calyces, solitary kidney, etc.) preventing the ability to direct a puncture laterally or render the subject stone free;
* Have participated in any other clinical trial within the last 3 months, and/or plans to participate in any other investigational or invasive clinical trial during this study;
* If female, breast-feeding, or if childbearing age, is not using contraception between screening and 90 days post-op;
* Subject has current or recent history of substance abuse (e.g. recreational drugs, narcotics, or alcohol) requiring intervention;
* Is a prisoner or ward of the state;
* Is unable to meet the treatment and follow up protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing percutaneous nephrolithotomy for treatment of their renal stone (s) total linear sum of 1.5 to 3cm cm in maximum dimension.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of successful renal access per access attempts | Procedure
  The proportion of successful renal access was compared to the renal access attempts (e.g. 100 success attempts/110 attempts).

SECONDARY OUTCOMES:
Location of Renal Access | Procedure
  The location of renal access was determined during the procedure. Location of access was defined as upper pole, mid pole, and lower pole.
Time to gain renal access | Procedure
  The time to gain renal access was defined as the time the ureteroscope enters the kidney to the time when the nephroscope enters the kidney
Total Procedure Time | Procedure
  The total procedure time is defined as the time when the cyso/urethroscope enters the urethra to the time time of skin closure.
Length of Post-Operative Hospital Stay | Day 0 to 3 Months Post-Operative
  The post-operative hospital length of stay range is defined from 0 days to longer than 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Whiles, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data collected during the study
Supporting Information: SAP, CSR
Time Frame: Following end of study
Access Criteria: Data may be requested by participating study investigators. The participating sites must have a data use agreement in place before requesting access to the data.

REFERENCES:
- [Background] Lee CL, Anderson JK, Monga M. Residency training in percutaneous renal access: does it affect urological practice? J Urol. 2004 Feb;171(2 Pt 1):592-5. doi: 10.1097/01.ju.0000104849.25168.6d. PMID 14713766
- [Background] Alotaibi KM. Retrograde nephrostomy access for percutaneous nephrolithotomy: a simple and safe technique. Urolithiasis. 2020 Apr;48(2):175-181. doi: 10.1007/s00240-019-01135-z. Epub 2019 Apr 29. PMID 31037404
- [Background] Kaler KS, Parkhomenko E, Lin CY, Valley ZA, Kim WK, Okhunov Z, Patel RM, Landman J. A New Twist on an Old Technique: Lawson Retrograde Endoscopic-Guided Nephrostomy Access for Percutaneous Nephrolithotomy in Prone Split-Leg Position. J Endourol Case Rep. 2018 Nov 29;4(1):190-194. doi: 10.1089/cren.2018.0073. eCollection 2018. PMID 30515460
- [Background] Wynberg JB, Paik LJ, Odom BD, Kruger M, Atalla CS. Body mass index predicts outcome of ureteroscopy-assisted retrograde nephrostomy for percutaneous nephrolithotomy. J Endourol. 2014 Sep;28(9):1071-7. doi: 10.1089/end.2014.0204. Epub 2014 Jun 12. PMID 24779944
- [Background] Sivalingam S, Al-Essawi T, Hosking D. Percutaneous nephrolithotomy with retrograde nephrostomy access: a forgotten technique revisited. J Urol. 2013 May;189(5):1753-6. doi: 10.1016/j.juro.2012.11.169. Epub 2012 Dec 3. PMID 23219545
- [Background] Al-Otaibi KM. Retrograde upper-pole calyceal access for percutaneous nephrolithotripsy of stones in the lower-pole calyx. Arab J Urol. 2012 Dec;10(4):353-7. doi: 10.1016/j.aju.2012.08.002. Epub 2012 Sep 23. PMID 26558049
- [Background] Kawahara T, Ito H, Terao H, Kato Y, Uemura H, Kubota Y, Matsuzaki J. Effectiveness of ureteroscopy-assisted retrograde nephrostomy (UARN) for percutaneous nephrolithotomy (PCNL). PLoS One. 2012;7(12):e52149. doi: 10.1371/journal.pone.0052149. Epub 2012 Dec 14. PMID 23251698
- [Background] Smiths Textbook of Endourology. 2007, BC Decker Publ. Ch. 15, Dr. D. Hosking - "Retrograde Nephrostomy", Pg. 117.
- [Background] Mokulis JA, Peretsman SJ. Retrograde percutaneous nephrolithotomy using the Lawson technique for management of complex nephrolithiasis. J Endourol. 1997 Apr;11(2):125-30. doi: 10.1089/end.1997.11.125. PMID 9107586
- [Background] Wong HY, Hinson JL, Griffith DP. Retrograde nephrostomy: advantages, disadvantages, and the learning curve. J Endourol. 1995 Dec;9(6):461-3. doi: 10.1089/end.1995.9.461. PMID 8775075
- [Background] Morrisseau PM, Trotter SJ. Retrograde percutaneous nephrolithotomy: urological treatment of a urological problem. J Urol. 1988 Jun;139(6):1163-5. doi: 10.1016/s0022-5347(17)42847-3. PMID 3373578
- [Background] Spirnak JP, Resnick MI. Retrograde percutaneous stone removal using modified Lawson technique. Urology. 1987 Dec;30(6):551-3. doi: 10.1016/0090-4295(87)90434-1. PMID 3686771
- [Background] Hunter PT, Hawkins IF, Finlayson B, Nanni G, Senior D. Hawkins-Hunter retrograde transcutaneous nephrostomy: a new technique. Urology. 1983 Dec;22(6):583-7. doi: 10.1016/0090-4295(83)90300-x. PMID 6649222
- [Background] Lawson RK, Murphy JB, Taylor AJ, Jacobs SC. Retrograde method for percutaneous access to kidney. Urology. 1983 Dec;22(6):580-2. doi: 10.1016/0090-4295(83)90299-6. PMID 6649221